CLINICAL TRIAL: NCT03976167
Title: Oxygen Administration During Bronchoscopy in Children, High Flow and Common Nasal Cannula: a Randomized Controled Trial
Brief Title: Comparison of Oxygen Adminstration by Nasal Cannula and High Flow Cannula During Bronchoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Son Espases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IB 3150/16 PI
Record Dates: First submitted 2019-05-30; First posted 2019-06-05 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Respiratory Disease
Keywords: Children; Desaturations; Bronchoscopy; Oxygen; High flow oxygen
MeSH Terms: conditions — Respiration Disorders | interventions — Oxygen Inhalation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Common nasal cannula (Active Comparator): Oxygen administration up to 4 liters according defined protocol
  Interventions: Device: Oxygen administration with Common nasal cannula
- High flow nasal cannula (Experimental): Oxygen administered with high flow nasal cannula according child weight and protocol designed for this study
  Interventions: Device: Oxygen administration with high flow nasal cannula, device Airvo2 Fisher and Pykel

INTERVENTIONS:
Device: Oxygen administration with Common nasal cannula — Oxygen administration during elective flexible bronchoscopy in children with high flow nasal cannula with inspired oxygen fraction 1.
  Arms: Common nasal cannula
Device: Oxygen administration with high flow nasal cannula, device Airvo2 Fisher and Pykel
  Arms: High flow nasal cannula

SUMMARY:
Randomized controled trial to compare oxygen desaturation during fiberoptic bronchoscopy using oxygen administered with nasal prongs and high flow nasal cannula. Drops in oxygen saturation are frequent during bronchoscopy and limit the procedure compromising patient security. The investigator's aim is to contribute to select better way of oxygen administration which could prevent desaturations during bronchoscopy in children.

ELIGIBILITY:
Inclusion Criteria:

* elective flexible bronchoscopy

Exclusion Criteria:

* admitted in Neonatal intensive care
* previous respiratory support: oxygen any device, non invasive or invasive ventilation
* patient who may benefit with continuous positive pressure during procedure

Ages: 29 Days to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2015-11-10 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Oxygen desaturation | Trough study completion, an average of 2 years
  Number of patients with Oxygen saturation under 94% during bronchoscopy

SECONDARY OUTCOMES:
Moderate oxygen desaturations | Trough study completion, an average of 2 years
  Number of patients with Oxygen saturation < 94% and > 90 %
Severe oxygen desaturations | Trough study completion, an average of 2 years
  Number of patients with Oxygen saturation< 90%
Tachypnea | Trough study completion, an average of 2 years
  Number of patients with Breath rate more than p95 fore age for more than 30 seconds
Apnea | Trough study completion, an average of 2 years
  Number of patients with Breath rate 0 for more than 20 seconds or recure intervention
Bradycardia | Trough study completion, an average of 2 years
  Number of patients with Heart rate less than p5 forte age for more than 20 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Artur sharluyan, MD, Principal Investigator — Ib-salut; Sebastian Sailer, MD, Study Director — Ib-salud; Francisco de Borja Osona Rodriguez, PhD, Study Chair — Ib-salud

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sharluyan A, Osona B, Frontera G, Brandstrup KB, Figuerola J, Sanz-Ruiz I, Salas A, Garrido B, Eva CG, Fernandez A, Pena-Zarza JA, Gil JA, Bover-Bauza C, Sailer S. High flow nasal cannula versus standard low flow nasal oxygen during flexible bronchoscopy in children: A randomized controlled trial. Pediatr Pulmonol. 2021 Dec;56(12):4001-4010. doi: 10.1002/ppul.25655. Epub 2021 Sep 10. PMID 34506689